CLINICAL TRIAL: NCT06689072
Title: Role of High Frequency Repetitive Transcranial Magnetic Stimulation in Management of Patients with Opioid Use Disorder in Upper Egypt
Brief Title: Role of High Frequency RTMS in Management of Opioid Use Disorder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sawy Alaa Sawy, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTMS in opioid patients in Egy; Assiut University (Other: Assiut University)
Record Dates: First submitted 2024-10-24; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Addiction; Opioid; RTMS
Keywords: Addiction; Opioid; rTMS; Egypt
MeSH Terms: conditions — Behavior, Addictive | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Group (Active Comparator): Participants diagnosed with Opioid use disorder
  Interventions: Other: rTMS
- Control Group (Sham Comparator): Participants who do not have Opioid use disoder
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Other: rTMS — To evaluate the role of repetitive Transcranial Magnetic Stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (DLPFC) in reducing pain, decreasing craving, alleviating withdrawal symptoms, lowering relapse rates, reducing impulsivity, and improving cognitive function in patients with Opioid Use Disorder
  Arms: Opioid Group
Behavioral: Psychotherapy — Using psychotherapy in opioid use disorder.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the role of repetitive Transcranial Magnetic Stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (DLPFC) in reducing pain, decreasing craving, alleviating withdrawal symptoms, lowering relapse rates, reducing impulsivity, and improving cognitive function in patients with Opioid Use Disorder, while also evaluating associated factors.

DETAILED DESCRIPTION:
Addiction is a complex, chronic brain condition influenced by genes and the environment that is characterized by substance use or compulsive actions that continue despite harmful consequences. For a long time, addiction meant an uncontrollable habit of using alcohol or other drugs as opioid. More recently, the concept of addiction has expanded to include behaviors, as well as substances, and even ordinary and necessary activities, such as exercise and eating.

Speaking of opioid addiction, Opioid addiction is a long-lasting (chronic) disease that can cause major health, social, and economic problems. Opioids are a class of drugs that act in the nervous system to produce feelings of pleasure and pain relief. Some opioids are legally prescribed by healthcare providers to manage severe and chronic pain. Commonly prescribed opioids include oxycodone, fentanyl, buprenorphine, methadone, oxymorphone, hydrocodone, codeine, and morphine. Some other opioids, such as heroin, are illegal drugs of abuse.

Opioid addiction is characterized by a powerful, compulsive urge to use opioid drugs, even when they are no longer required medically. Opioids have a high potential for causing addiction in some people, even when the medications are prescribed appropriately and taken as directed. Many prescription opioids are misused or diverted to others. Individuals who become addicted may prioritize getting and using these drugs over other activities in their lives, often negatively impacting their professional and personal relationships. It is unknown why some people are more likely to become addicted than others.

ELIGIBILITY:
Inclusion criteria:

* Male
* Age 18- 40
* Opioid use disorder

Exclusion criteria:

* Individuals with mental disorders (such as primary psychosis, schizophrenia, mental retardation, and brain damage induced mental disorder),
* History of epilepsy
* History of cardiovascular complications.
* History of contraindications to TMS (e.g. metal implants in the head).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Role of rTMS in managing opioid use disorders using multiple scales | 2 years
  To evaluate the role of repetitive Transcranial Magnetic Stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (DLPFC) in reducing pain in patients with Opioid Use Disorder by using BRIEF PAIN INVENTORY (SHORT FORM) scale.
RTMS in managing opioid use disorder in Upper Egypt | 2 years
  Repetitive Transcranial Magnetic Stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (DLPFC) in reducing craving in opioid use disorder patient using Brief Substance Craving Scale.
RTMS in managing opioid use disorder in Upper Egypt | 2 years
  Repetitive Transcranial Magnetic Stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (DLPFC) in improving cognition using Montreal Cognitive Assessment (MoCA) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Because I have not take the permission from supper visors yet

REFERENCES:
- [Background] Yang S, Chang MC. Effect of Repetitive Transcranial Magnetic Stimulation on Pain Management: A Systematic Narrative Review. Front Neurol. 2020 Feb 18;11:114. doi: 10.3389/fneur.2020.00114. eCollection 2020. PMID 32132973
- [Background] Addolorato G, Antonelli M, Cocciolillo F, Vassallo GA, Tarli C, Sestito L, Mirijello A, Ferrulli A, Pizzuto DA, Camardese G, Miceli A, Diana M, Giordano A, Gasbarrini A, Di Giuda D. Deep Transcranial Magnetic Stimulation of the Dorsolateral Prefrontal Cortex in Alcohol Use Disorder Patients: Effects on Dopamine Transporter Availability and Alcohol Intake. Eur Neuropsychopharmacol. 2017 May;27(5):450-461. doi: 10.1016/j.euroneuro.2017.03.008. Epub 2017 Apr 6. PMID 28390775
- [Background] Liu X, Zhao X, Liu T, Liu Q, Tang L, Zhang H, Luo W, Daskalakis ZJ, Yuan TF. The effects of repetitive transcranial magnetic stimulation on cue-induced craving in male patients with heroin use disorder. EBioMedicine. 2020 Jun;56:102809. doi: 10.1016/j.ebiom.2020.102809. Epub 2020 Jun 5. PMID 32512513
- [Background] Tsai TY, Wang TY, Liu YC, Lee PW, Chang WH, Lu TH, Tseng HH, Lee SY, Chang YH, Yang Y, Chen PS, Chen KC, Yang YK, Lu RB. Add-on repetitive transcranial magnetic stimulation in patients with opioid use disorder undergoing methadone maintenance therapy. Am J Drug Alcohol Abuse. 2021 May 4;47(3):330-343. doi: 10.1080/00952990.2020.1849247. Epub 2021 Jan 10. PMID 33426970
- [Background] Imperatore JP, McCalley DM, Borckardt JJ, Brady KT, Hanlon CA. Non-invasive brain stimulation as a tool to decrease chronic pain in current opiate users: A parametric evaluation of two promising cortical targets. Drug Alcohol Depend. 2021 Jan 1;218:108409. doi: 10.1016/j.drugalcdep.2020.108409. Epub 2020 Nov 23. PMID 33250384